CLINICAL TRIAL: NCT03330015
Title: Patient's Experience and Choice Between Investigations for Endometrial Cancer in Postmenopausal Bleeding
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fung Wen Ying Linda, Associate Consultant, Chinese University of Hong Kong
Other Study IDs: CREC 2015.437
Record Dates: First submitted 2017-10-25; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-09

CONDITIONS: Endometrial Cancer; Postmenopausal Bleeding
Keywords: postmenopausal bleeding; endometrial cancer; Patient's experience; Patient's choice
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endometrial cancer is the most common malignancy of the female genital tract in Hong Kong. The aim in the evaluation of PMB is to exclude underlying malignancy. Endometrial thickness (ET) measured by transvaginal ultrasound scanning (TVS) and endometrial biopsy or sampling (ES) has been recommended as the first-line investigation. From a study between 2002-2013 in the One-stop PMB clinic, investigators found that ET was able to identify women with endometrial cancer with the sensitivity at 3mm, 4mm, and 5mm, the current levels recommended in professional guidelines, being 97.0%, 94.1%, and 93.5% respectively. However, little is known about the level of patient's acceptance of the false negative rate and how patient would trade residual risk with more invasive test. There is also a lack of study on the experience of women during the management pathway especially the level of anxiety before and after investigations and the pain experienced from the investigations offered. The current study aim to study the level of false negative rate accepted by women for the investigation of PMB and the level of anxiety and pain experienced during the investigation pathway.

DETAILED DESCRIPTION:
Endometrial cancer is the most common malignancy of the female genital tract in Hong Kong. It is estimated that around 10% of women experience postmenopausal bleeding. Around 90% of women with endometrial cancer initially presented with postmenopausal bleeding (PMB). The aim in the evaluation of PMB is to exclude underlying malignancy. Clinical tests to evaluate the endometrium include transvaginal ultrasound scanning (TVS) to measure endometrial thickness (ET), endometrial biopsy or sampling (ES), saline infusion sonography, and hysteroscopy. TVS ET or ES has been recommended as the first-line investigation.

There are, however, different ET cut-off values recommended by various professional groups. From a study between 2002-2013 in the One-stop PMB clinic, investigators found that ET was able to identify women with endometrial cancer with the sensitivity at 3mm, 4mm, and 5mm, the current levels recommended in professional guidelines, being 97.0%, 94.1%, and 93.5% respectively.

Although clinical management guidelines and accuracy data are available, little is known about the level of patient's acceptance of the false negative rate and how patient would trade residual risk with more invasive test. There is also a lack of study on the experience of women during the management pathway especially the level of anxiety before and after investigations and the pain experience from the investigations offered. There is only one study identified from the literature which suggested high levels of anxiety in women who experienced PMB.

There is a dedicated Postmenopausal Bleeding Clinic for the one-stop evaluation for PMB in Hong Kong and investigators receive referrals from other centers in Hong Kong. It is a tertiary-care university institution with two affiliated hospitals.

All patients who are new referrals for the symptom of PMB will be invited to participate in the study. Informed consent form will be obtained from all patients participating in the study. Patients will be asked to read written information on postmenopausal bleeding including the risk of endometrial cancer and investigation options including TVS ET, hysteroscopy and ES. The information will be focused on the detection rate and procedure-related risk. The interviewer will specify that 1) hysteroscopy and ES will be considered to offer 100% detection rate but there is procedure related risks including pain, bleeding, infection, uterine perforation because entrance into the uterine cavity is required 2) TVS ET do not require entry into uterine cavity but the detection rate is not 100%. Then patients will undergo a structured interview by an interviewer using the standard gamble technique.

In the standard gamble test, patients will be asked to choose from a guaranteed outcome (e.g. being blind for the rest of their life), or whether patients would prefer an alternative state with some chance of a worst outcome (e.g. dying, "1-p") and a complementary chance of an ideal outcome (e.g. continue to live healthily, "p"). The risks of the two situations will be varied until the patient is unable to decide either of the two options. This allows quantitative comparison of the health states, which allow us to understand the decision -making process of the patient. The interviewer will use blindness, death and healthy life to ensure the patient understand the standard gamble method. The participant will be asked to make a decision starting with a probability of 100%, which will then be reduced in steps of 10% until it reach 10% after which it will be decreased at 1% interval until 2% and thereafter at 0.1% interval, until the participant is not unable to make a choice between the two options.

Then the exercise will be repeated to test the preferences towards the investigations for PMB. The patient will be asked to choose between one of the tests (1) TVS ET (2) hysteroscopy with ES. In order to determine the level of acceptance of false negative rate using TVS ET, the assumed detection rate of the test will be quoted as 75% and increase in steps in 5% interval until it reach 90%, then increase at 1% interval until it reach 98%, and then at 0.1% interval until it reach 99.9%.

The anxiety level will be assessed by the Full form State-Anxiety scale. Since anxiety may be affected by the anticipated pain associated with each investigation. Patient's idea about the potential pain which will experience from the different investigations (TVS ET, hysteroscopy, ES) will be rated by a visual analogue scale from 0-10.

The patient will then enter the consultation room and have the PMB assessment. After the consultation, the patient will be interviewed again. The standard gamble and anxiety level will be assessed again to determine if the actual experience after the PMB assessments changed the patients' choice. The actual VAS score on the investigations received will be recorded. The patient will then be asked to complete the same anxiety questionnaire 3 months from the consultation and return by the return envelops provided.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal woman
* referrals for the symptom of PMB

Exclusion Criteria:

* dementia
* mental retardation

Ages: 40 Years to 69 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Our center provides a dedicated Postmenopausal Bleeding Clinic for the one-stop evaluation for PMB in Hong Kong and we receive referrals from other centers in Hong Kong. Our center is a tertiary-care university institution with two affiliated hospitals.All patients who are new referrals for the symptom of PMB will be invited to participate in the study. A woman is considered to have PMB if there is occurrence of bleeding after one completed year of amenorrhoea.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
The level of acceptance of false negative rate using TVS ET | Baseline
  The level of acceptance of false negative rate using endometrial thickness assessed by transvaginal ultrasound scanning to identify endometrial cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Ying Fung, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong